CLINICAL TRIAL: NCT03215628
Title: Quantifizierung Der Hirnperfusion Während Kinderherzchirurgischer Operationen Durch Transkraniellen Kontrastmittelverstärkten Ultraschall
Brief Title: Quantification of Cerebral Perfusion by Contrast-enhanced Ultrasound During Neonatal Heart Surgery
Acronym: TCEUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20_17B
Record Dates: First submitted 2017-07-04; First posted 2017-07-12 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2020-11

CONDITIONS: Heart Defects, Congenital
Keywords: CEUS; TCEUS; contrast enhanced ultrasound; perfusion; cerebral perfusion; sulphur hexafluoride; SonoVue
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A - TCEUS with HLM (Active Comparator): General neonatal cardiac surgery with HLM (art. switch, aortopulmonary shunts)
  Interventions: Diagnostic Test: TCEUS
- Group B - TCEUS with HLM (Experimental): Surgery of the aortic arc
  Interventions: Diagnostic Test: TCEUS
- Group C - TCEUS without HLM (Active Comparator): Neonatal cardiac surgery without HLM
  Interventions: Diagnostic Test: TCEUS

INTERVENTIONS:
Diagnostic Test: TCEUS — Intravenous sulphur hexafluoride microbubbles
  Other Names: Transcranial contrast-enhanced ultrasound

SUMMARY:
Transcranial contrast-enhanced ultrasound for evaluation of cerebral blood flow during pediatric cardiac surgery. This study is aimed as a feasibility study prior to conducting a lager prospective clinical trial including neurologic and developmental outcome measures.

DETAILED DESCRIPTION:
The cerebral perfusion of infants with congenital heart defects is a critical determinant during cardiac surgery. The majority of these interventions is performed during deep or moderate hypothermia (25-32°C) with reduced blood flow of the heart-lung-machine (HLM). Assuming a symmetrical anatomy of the cerebral arteries (C. Willisii) a single vessel (T. brachiocephalicus) is then supplying the cerebral blood flow. Using contrast-enhanced ultrasound the cerebral blood flow will be assessed during cardiac surgery interventions.

ELIGIBILITY:
Inclusion Criteria:

* Neonates and infants ≤ 4 month (open fontanelle)
* Proper ultrasound conditions/window
* Appropriate general and neurologic state of health
* Written consent of both parents/guardians
* Availability of trained sonographer (medical doctor)

Exclusion Criteria:

* Absence of trained sonographer (medical doctor)
* Intolerance against SonoVue® (bzw. sulphur hexafluoride)
* Missing signed consent
* Reduced or inappropriate general and neurologic state of health
* Preexisting cerebral injury

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Time-To-Peak (TTP) | Intraoperative (Directly after start of surgical intervention (T1) vs. Directly before end of intervention (T5))
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software
Mean-Transit-Time (MTT) | Intraoperative (Directly after start of surgical intervention (T1) vs. Directly before end of intervention (T5))
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software
Maximum Intensity (MI) | Intraoperative (Directly after start of surgical intervention (T1) vs. Directly before end of intervention (T5))
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software
Relative Blood Volume (RBV) | Intraoperative (Directly after start of surgical intervention (T1) vs. Directly before end of intervention (T5))
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software
Relative Blood Flow (RBF) | Intraoperative (Directly after start of surgical intervention (T1) vs. Directly before end of intervention (T5))
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software

SECONDARY OUTCOMES:
Time-To-Peak (TTP) | Directly after start of surgical intervention (T1) vs. Directly after full flow of HLM at 37°C (T2)
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software
Time-To-Peak (TTP) | Directly after start of surgical intervention (T1) vs. Directly after full flow of HLM at 25-28°C/hypothermia (T3)
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software
Time-To-Peak (TTP) | Directly after start of surgical intervention (T1) vs. Directly after low flow of HLM at 25-28°C/hypothermia (T4)
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software
Mean-Transit-Time (MTT) | Directly after start of surgical intervention (T1) vs. Directly after full flow of HLM at 37°C (T2)
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software
Mean-Transit-Time (MTT) | Directly after start of surgical intervention (T1) vs. Directly after full flow of HLM at 25-28°C/hypothermia (T3)
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software
Mean-Transit-Time (MTT) | Directly after start of surgical intervention (T1) vs. Directly after low flow of HLM at 25-28°C/hypothermia (T4)
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software
Maximum Intensity (MI) | Directly after start of surgical intervention (T1) vs. Directly after full flow of HLM at 37°C (T2)
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software
Maximum Intensity (MI) | Directly after start of surgical intervention (T1) vs. Directly after full flow of HLM at 25-28°C/hypothermia (T3)
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software
Maximum Intensity (MI) | Directly after start of surgical intervention (T1) vs. Directly after low flow of HLM at 25-28°C/hypothermia (T4)
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software
Relative Blood Volume (RBV) | Directly after start of surgical intervention (T1) vs. Directly after full flow of HLM at 37°C (T2)
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software
Relative Blood Volume (RBV) | Directly after start of surgical intervention (T1) vs. Directly after full flow of HLM at 25-28°C/hypothermia (T3)
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software
Relative Blood Volume (RBV) | Directly after start of surgical intervention (T1) vs. Directly after low flow of HLM at 25-28°C/hypothermia (T4)
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software
Relative Blood Flow (RBF) | Directly after start of surgical intervention (T1) vs. Directly after full flow of HLM at 37°C (T2)
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software
Relative Blood Flow (RBF) | Directly after start of surgical intervention (T1) vs. Directly after full flow of HLM at 25-28°C/hypothermia (T3)
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software
Relative Blood Flow (RBF) | Directly after start of surgical intervention (T1) vs. Directly after low flow of HLM at 25-28°C/hypothermia (T4)
  Relative/percentage difference of cerebral perfusion by TCEUS-based quantification using VueBox(R) software

CONTACTS AND LOCATIONS:
Overall Officials: André Rüffer, MD, Principal Investigator — University Hospital Erlangen, Department of Pediatric Cardiac Surgery; Jörg Jüngert, MD, Principal Investigator — University Hospital Erlangen, Department of Pediatrics
Locations (1):
- University Hospital of Erlangen-Nürnberg, Department of Pediatric Cardiac Surgery, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Knieling F, Cesnjevar R, Regensburger AP, Wagner AL, Purbojo A, Dittrich S, Munch F, Neubert A, Woelfle J, Jungert J, Ruffer A. Transfontanellar Contrast-enhanced US for Intraoperative Imaging of Cerebral Perfusion during Neonatal Arterial Switch Operation. Radiology. 2022 Jul;304(1):164-173. doi: 10.1148/radiol.212044. Epub 2022 Apr 5. PMID 35380495
- [Derived] Ruffer A, Knieling F, Cesnjevar R, Regensburger A, Purbojo A, Dittrich S, Munch F, Wolfle J, Jungert J. Equal cerebral perfusion during extended aortic coarctation repair. Eur J Cardiothorac Surg. 2022 Jan 24;61(2):299-306. doi: 10.1093/ejcts/ezab415. PMID 34718510